CLINICAL TRIAL: NCT06187220
Title: Effect of Therapeutic Plasma Exchange on Liver Transplantation-free Survival in Amanita Toxin-induced Acute Liver Failure - a Multicenter Retrospective Study Over 10 Years
Brief Title: Plasma Exchange for Amanita Toxin-induced Acute Liver Failure
Acronym: Amanita-Pex
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Stahl, Klaus Dr., PD Dr. Klaus Stahl, PD Dr. Richard Taubert, Dr. Bahar Nalbant, Hannover Medical School
Other Study IDs: Amanita-Pex
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Liver Failure
Keywords: Liver Failure; Amanita Toxin; Plasmapheresis; Liver Transplantation
MeSH Terms: conditions — Liver Failure, Acute; Liver Failure | interventions — Plasma Exchange

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Therapeutic Plasma Exchange (PEX): Patients receiving in addition to Standard Medical Therapy (SMT) at least one treatment with Therapeutic Plasma Exchange (PEX)
  Interventions: Device: Therapeutic Plasma Exchange (PEX)
- Standard Medical Therapy (SMT): Patients receiving only Standard Medical Therapy (SMT) of Amanita Toxin associated acute liver failure, including intensive care support (invasive ventilation, vasopressors, renal replacement therapy), silibinin and n-acetylcystein. Included in this group are also patients receiving albumine dialysis or other extracorporeal liver assist therapies excluding therapeutic plasma exchange.

INTERVENTIONS:
Device: Therapeutic Plasma Exchange (PEX) — Therapeutic plasma exchange with treatment sessions >=1 replacing varying fractions of patient´s whole plasma with healthy donor plasma
  Groups: Therapeutic Plasma Exchange (PEX)

SUMMARY:
Retrospective evaluation of the value of additive therapeutic plasma exchange (PEX) compared to standard medical therapy (SMT) in Amanita toxin-associated acute liver failure in children and adolescents within the last 10 years at a international group of liver transplant centers.

DETAILED DESCRIPTION:
Amanita toxin-associated acute liver failure is a life-threatening condition that can often lead to the need for an emergency liver transplantation. The disease may also be fatal, particularly in patients who are not eligible for a liver transplant due to advanced age or corresponding comorbidities.

Therapeutic plasma exchange treatment has been shown to significantly improve patient survival in other cases of acute liver failure and has since become standard treatment for acute liver failure in many, but not all, liver transplant centers. However, no patients with Amanita toxin-associated acute liver failure were included in these cohorts.

The hypothesis of the planned study is that an additive therapeutic plasma exchange treatment (PEX) can improve liver transplantation-free survival in these patients compared to standard medical therapy (SMT) alone. Since the therapy procedure in different transplant centers in differs with regard to the use of therapeutic plasma exchange, we are therefore planning a multicenter retrospective comparison of PEX with SMT with regard to transplant-free survival and other clinical endpoints. For this very small cohort of patients with acute liver failure, which also varies in frequency depending on the season and weather conditions, there will certainly never be a sufficiently powered randomized and controlled study. This analysis may change the standard procedure for patients with Amanita toxin-associated acute liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Acute liver failure (presence of hepatic encephalopathy of grade I or higher and a coagulopathy with an INR > 1.5)
* Amanita Toxin related acute liver failure

Exclusion Criteria:

* Acute liver failure of other reason than Amanita Toxin
* Amanita Toxin associated Hepatitis or severe hepatitis without fulfilling the criteria of acute liver failure

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Amanita toxin related acute liver failure, both adult and pediatric
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Liver Transplant free Survival | until day 28 from initial diagnosis of acute liver failure
  Survival and free of liver transplantation until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)

SECONDARY OUTCOMES:
Overall Survival | until day 28 from initial diagnosis of acute liver failure
  Survival until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with International normalized ratio (INR) > 1.5)
Liver transplantation | until day 28 from initial diagnosis of acute liver failure
  Liver transplantation until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
High urgency (HU) listing for liver transplantation | until day 28 from initial diagnosis of acute liver failure
  Initiated high urgency listing for liver transplantation until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
Acute kidney injury (AKI) and max. grade of AKI (I-III) | until day 28 from initial diagnosis of acute liver failure
  Acute kidney injury and max. grade of AKI (I-III) until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
Renal Replacement Therapy (RRT) | until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
  Initiated renal replacement therapy until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
Vasopressor therapy | until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
  Initiated vasopressor therapy until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
Invasive ventilation | until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
  Initiated invasive ventilation until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
Maximum grade of hepatic encephalopathy (HE) | until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)
  Maximum grade of hepatic encephalopathy (HE) until day 28 from initial diagnosis of acute liver failure (encephalopathy of any grade and coagulopathy with INR > 1.5)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Stahl, MD, Principal Investigator — Hannover Medical School, Hannover Germany; Richard Taubert, MD, Principal Investigator — Hannover Medical School, Hannover Germany
Locations (6):
- Germany (2):
  - University Hospital Aachen (RWTH), Aachen
  - Hannover Medical School, Hanover
- ASST Ospedale Papa Giovanni XXIII, Bergamo, Italy
- INCMNSZ, Mexico City, Mexico
- Curry Cabral Hospital, Lisbon, Portugal
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share on reasonable request

REFERENCES:
- [Background] Stahl K, Hadem J, Schneider A, Manns MP, Wiesner O, Schmidt BMW, Hoeper MM, Busch M, David S. Therapeutic plasma exchange in acute liver failure. J Clin Apher. 2019 Oct;34(5):589-597. doi: 10.1002/jca.21737. Epub 2019 Jul 26. PMID 31348553
- [Background] Stahl K, Bode C, David S. Bridging patients with acute-on-chronic liver failure for transplantation: plasma exchange to stabilize multiorgan failure? Intensive Care Med. 2023 Jul;49(7):890-891. doi: 10.1007/s00134-023-07092-x. Epub 2023 May 13. No abstract available. PMID 37178148
- [Background] Stahl K, Busch M, Fuge J, Schneider A, Manns MP, Seeliger B, Schmidt JJ, Wiesner O, Schmidt BMW, Taubert R, Vondran FWR, Hoeper MM, David S. Therapeutic plasma exchange in acute on chronic liver failure. J Clin Apher. 2020 Aug;35(4):316-327. doi: 10.1002/jca.21799. Epub 2020 Jun 24. PMID 32583446